CLINICAL TRIAL: NCT04642014
Title: A Multi-centre, 18-months, Single-group Study of Application of Convalescent Plasma in the Treatment of SARS CoV-2 Disease (COVID-19) With Metabolomic and Laboratory Evaluation of Plasma Therapy Effectiveness
Brief Title: Application of Convalescent Plasma in the Treatment of SARS CoV-2 Disease (COVID-19) With Evaluation of Therapy Effectiveness
Acronym: EPIC-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The main reasons for the premature termination of the study are the inability to reliably assess the effectiveness of therapy due to the emergence of new variants of SARS-CoV-2 and reports of the lack of benefits of using plasma in previous studies.
Sponsor: Wroclaw Medical University (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020.ABM.COVID19.0005
Record Dates: First submitted 2020-11-23; First posted 2020-11-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2020-11

CONDITIONS: COVID-19 Convalescent Plasma Treatment
MeSH Terms: interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: The study is going to recruit 300 convalescent plasma donors and 200 recipients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized patients with SARS CoV-2 infection (Experimental): Hospitalized patients with SARS CoV-2 infection will receive an anti SARS-CoV-2 convalescent plasma
  Interventions: Biological: COVID-19 convalescent plasma treatment

INTERVENTIONS:
Biological: COVID-19 convalescent plasma treatment — The donor's blood will be collected after four weeks post-onset of illness. 600 ml ABO-compatible plasma sample will be harvested during apheresis from each donor and each sample will be divided and stored as 200 mL aliquots.
  Patients who meet the criteria receive one dose (200 mL) of ABO compatible inactivated convalescent plasma with a confirmed neutralization activity.

SUMMARY:
A Multi-centre, 18-months, Single-group Study of Application of Convalescent Plasma in the Treatment of SARS CoV-2 Disease (COVID-19) With Metabolomic and Laboratory Evaluation of Plasma Therapy Effectiveness.

DETAILED DESCRIPTION:
The trial is designed as multi-centre, non-randomized, single-group with a primary endpoint of death of convalescent plasma recipient in twenty eight days. We are planning to recruit 300 donor patients who recovered from COVID-19 and who offer to take part in an experiment based on the informed consent form. The recovery criteria involve body temperature normalization for more than 3 days, resolution of respiratory tract symptoms, and two consecutively negative results of SARS-CoV-2 RT-PCR assay test. The donor's blood will be collected after four weeks post-onset of illness. 600 ml ABO-compatible plasma sample will be harvested during apheresis from each donor and each sample will be divided and stored as 200 mL aliquots. The plasma recipients are adult patients diagnosed with COVID-19 according to the WHO Interim Guidance with confirmation by real-time RT-PCR assay The inclusion criteria to receive plasma assume to meet at least one of following : respiratory distress with tachypnoe ≥30 breaths per minute, oxygen level less than 94% in resting-state, partial pressure of oxygen (PO2) ≤ 80 mmHg. Patients who meet the criteria receive one dose (200 mL) of ABO compatible inactivated convalescent plasma with a confirmed neutralization activity. The recipient are going to undergo detailed clinical evaluation along with the assessment of biochemical parameters, complete blood count and inflammation indicators. The study involves a comprehensive assessment of the serological response of patients with different course of SARS-Cov-2 infection, as well as an analysis of the impact of the level of antibodies in the donor's plasma on the clinical response in patients with COVID-19. In addition, a comprehensive metabolomic analysis of donor and recipient blood was planned to identify prognostic and predictive factors. The endpoints include the safety of convalescents plasma transfusion, as well as the improvement of clinical symptoms and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

Donors:

1. Age >18 and <65 years
2. Confirmed previous SARS CoV-2 infection
3. Signed informed consent to participate in this clinical trial, to donate plasma and to store the specimen for future testing.
4. At least 28 days from the end of isolation or resolution of symptoms of infection
5. Male donors, or female donors who have not been pregnant, or female donors who have been pregnant tested negative for HLA antibodies
6. Individuals who meet all regular voluntary donor eligibility requirements

Recipiants:

1. Signed informed consent to participate in this clinical trial.
2. Confirmed previous SARS CoV-2 infection
3. Respiratory distress with tachypnoe ≥30 breaths per minute,
4. Oxygen level less than 94% in resting-state,
5. Partial pressure of oxygen (PO2) ≤ 80 mmHg

Exclusion Criteria:

Donors:

1. Age : <18 or >65 years
2. Female subjects who are pregnant
3. HIV1,2 hepatitis B,C or syphilis infection
4. Donors ineligible for regular voluntary blood donation

Recipiants:

1. No informed consent to participate in the study
2. Patients with a history of plasma hypersensitivity, including anaphylactic shock in previous transfusions, allergic reactions to citrate or primary IgA deficiency
3. Patients with symptoms of severe multi-organ failure
4. Patients with known allergic reactions to chemical compounds used or generated in the procedure of inactivation of pathogens
5. Patients with active thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Death, for any reason | 28 days after transfusion
  Death, for any reason

SECONDARY OUTCOMES:
For patients with respiratory support, the time to take one's own breath (extubation) | 28 days after transfusion
  For patients with respiratory support, the time to take one's own breath (extubation)
Stay in the intensive care unit (ICU) | 28 days after transfusion
  Stay in the intensive care unit (ICU)
Time to disconnect CPAP respiratory support | 28 days after transfusion
  Time to disconnect CPAP respiratory support
Time to elimination of SARS-Cov-2 (RT-PCR) | 28 days after transfusion
  Time to elimination of SARS-Cov-2 (RT-PCR)
Time to serological response (anti-SARS-COv-2 antibodies) | 3, 7, 28 days after transfusion
  Time to serological response (anti-SARS-COv-2 antibodies)

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Rajendran K, Krishnasamy N, Rangarajan J, Rathinam J, Natarajan M, Ramachandran A. Convalescent plasma transfusion for the treatment of COVID-19: Systematic review. J Med Virol. 2020 Sep;92(9):1475-1483. doi: 10.1002/jmv.25961. Epub 2020 May 12. PMID 32356910
- [Background] Li L, Zhang W, Hu Y, Tong X, Zheng S, Yang J, Kong Y, Ren L, Wei Q, Mei H, Hu C, Tao C, Yang R, Wang J, Yu Y, Guo Y, Wu X, Xu Z, Zeng L, Xiong N, Chen L, Wang J, Man N, Liu Y, Xu H, Deng E, Zhang X, Li C, Wang C, Su S, Zhang L, Wang J, Wu Y, Liu Z. Effect of Convalescent Plasma Therapy on Time to Clinical Improvement in Patients With Severe and Life-threatening COVID-19: A Randomized Clinical Trial. JAMA. 2020 Aug 4;324(5):460-470. doi: 10.1001/jama.2020.10044. PMID 32492084
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Ye M, Fu D, Ren Y, Wang F, Wang D, Zhang F, Xia X, Lv T. Treatment with convalescent plasma for COVID-19 patients in Wuhan, China. J Med Virol. 2020 Oct;92(10):1890-1901. doi: 10.1002/jmv.25882. Epub 2020 Jun 29. PMID 32293713
- [Background] Yigenoglu TN, Hacibekiroglu T, Berber I, Dal MS, Basturk A, Namdaroglu S, Korkmaz S, Ulas T, Dal T, Erkurt MA, Turgut B, Altuntas F. Convalescent plasma therapy in patients with COVID-19. J Clin Apher. 2020 Aug;35(4):367-373. doi: 10.1002/jca.21806. Epub 2020 Jul 9. PMID 32643200
- [Background] Joyner MJ, Wright RS, Fairweather D, Senefeld JW, Bruno KA, Klassen SA, Carter RE, Klompas AM, Wiggins CC, Shepherd JR, Rea RF, Whelan ER, Clayburn AJ, Spiegel MR, Johnson PW, Lesser ER, Baker SE, Larson KF, Ripoll JG, Andersen KJ, Hodge DO, Kunze KL, Buras MR, Vogt MN, Herasevich V, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Van Buskirk CM, Winters JL, Stubbs JR, Paneth NS, Verdun NC, Marks P, Casadevall A. Early safety indicators of COVID-19 convalescent plasma in 5000 patients. J Clin Invest. 2020 Sep 1;130(9):4791-4797. doi: 10.1172/JCI140200. PMID 32525844